CLINICAL TRIAL: NCT05214794
Title: An Open-label, Phase 2 Study to Assess the Efficacy and Safety of Nemolizumab in Subjects With Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M525101-21
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — nemolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nemolizumab (Experimental)
  Interventions: Drug: nemolizumab

INTERVENTIONS:
Drug: nemolizumab — nemolizumab will be administered subcutaneous injection

SUMMARY:
To evaluate the efficacy of nemolizumab in systemic sclerosis patients. To evaluate also the safety and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Sclerosis according to American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) 2013 criteria
* Systemic Sclerosis patients with moderate to sever skin sclerosis

Exclusion Criteria:

* Patients witg a disease considered inappropriate for participation in clinical trials, such as serious cardiac / hepatic / renal / pulmonary / hematologic disease
* Patients with a diseases that could interfere with assessment of Systemic Scleorosis
* Patients with body weight less than 30.0kg
* Pregnant or lactating women.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in modified Rodnan Skin Score (mRSS) at Week 24 | Baseline and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Ayumi Yoshizaki, MD, PhD, Principal Investigator — Tokyo University
Locations (1):
- The University of Tokyo Hospital, Tokyo, Japan